CLINICAL TRIAL: NCT03705572
Title: A Randomised, Double-blind, Parallel Groups, Placebo-controlled 6 Week Human Intervention Study Investigating the Effect of a Phospholipid Drink on Cognitive Performance in 6-8 Year Old School Children
Brief Title: Intervention Study Investigating the Effect of a Phospholipid Drink on Cognitive Performance in 6-8 Year Old School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Arla02
Record Dates: First submitted 2016-07-07; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Milk; Lacprodan PL20; Glycerophospholipids; Cognition
MeSH Terms: interventions — lacprodan PL-20

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement: Phospholipid drink. (Active Comparator): Participant in an intervention parallel group consumed a drink with added phospholipids (Lacprodan PL20).
  Interventions: Dietary Supplement: Lacprodan PL20
- Dietary Supplement: Placebo milk drink. (Placebo Comparator): Participant in an intervention parallel group consumed a drink without added phospholipids.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lacprodan PL20 — Milk protein concentrate that is high in phospholipid content (min 16%).
  Arms: Dietary Supplement: Phospholipid drink.
Other: Placebo — Placebo milk drink.
  Arms: Dietary Supplement: Placebo milk drink.

SUMMARY:
Six week RCT intervention on the effects of phospholipid containing milk drink vs. placebo milk drink on cognitive performance in 6-8 year old school children.

DETAILED DESCRIPTION:
A randomised, double blind, placebo controlled study with parallel groups investigating a 6 week intervention in 6-8 year old school children of phospholipid containing milk drink vs. placebo milk drink. Participants were familiarised with the test battery and IQ (Wechsler abbreviated scale of intelligence) and colour blindness (Ishihara test) measurements were taken prior to the intervention. Milk drink taste testing and milk preference selection was also carried out prior to the intervention. The test battery was administered at baseline (week 0), midpoint (week 3) and endpoint (week 6), and the milk intervention was given Monday - Friday at school shortly before their mid-morning break over a 6 week period. This study design, including both the test days and morning milk supplementation, was intended to emulate the children's normal routine as far as possible. The milk drink was a supplement to the children's usual diet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 6-8 years.
* Willingness to consume milk drinks during the study determined by a score of >5 on a taste testing Likert scale for at least one flavour of the milk drinks.
* Ability to follow verbal and simple written instructions in English.
* Normal vision, with appropriate corrective lenses if required.
* Ability to understand cognitive testing instructions and responding requirements.

Exclusion Criteria:

* Poor general health.
* Colour blindness.
* Behavioural difficulties or attention disorders (e.g. Attention Deficit Hyperactivity Disorder).
* Learning disabilities that interfere with the ability to understand written or verbal communications.
* Inability to understand the objective of the cognitive tests, or carry out the tests.
* Any food allergies or intolerances (e.g. lactose intolerance).
* Acute illness, or feelings of unwell, within the week prior to testing.
* Current administration of any psychotropic medication or supplementation in the month prior to testing, or during testing.
* Hearing impairment that precludes the ability to follow verbal instructions.
* Children already receiving milk at school unless parents are willing to substitute current milk with the study milk.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Rivermead Behavioural Memory Test for Children (RBMT-C) change from baseline | Week 0, week 3 & week 6
  Test of immediate and delayed verbal memory recall.

SECONDARY OUTCOMES:
Motor Screening Task (CANTAB suite) change from baseline | Week 0, week 3 & week 6
  To identify motor impairment. Dependent variables: reaction time for each trial and distance from cross.
Spatial Recognition Memory (CANTAB suite) change from baseline | Week 0, week 3 & week 6
  Dependent variables: number of correct trials and reaction time for each trial.
Spatial Span (CANTAB suite) change from baseline | Week 0, week 3 & week 6
  Dependent variables: highest span reached, number of correct responses, number of incorrect responses and reaction time for each trial.
Reaction time (CANTAB suite) change from baseline | Week 0, week 3 & week 6
  Dependent variables: mental reaction time and movement time for each trial, number of correct responses, number of incorrect responses and number of invalid responses. Two parts to the task included simple, one response option, and choice, 5 response options.
Subjective mood questionnaire change from baseline | Week 0, week 3 & week 6
  Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Dye, PhD, Principal Investigator — Professor of Nutrition & Behaviour; Lead for Strategic Development.; Clare Lawton, PhD, Principal Investigator — Associate Professor of Nutrition & Behaviour.

IPD SHARING:
Plan to Share IPD: No